CLINICAL TRIAL: NCT05227924
Title: Safety and Performance Assessment of the SYMBOL Range of Medical Devices in Patients Underlying Total Hip Arthroplasty
Status: Recruiting | Type: Observational
Sponsor: Dedienne Sante S.A.S. (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: PMCF_SYMBOL_01
Record Dates: First submitted 2021-12-02; First posted 2022-02-08 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Degenerative Hip Joint Disease; Post-traumatic Osteoarthritis; Hip Arthritis; Femoral Neck Fractures; Avascular Necrosis of the Femoral Head; Failure of Prosthetic Joint Implant
MeSH Terms: conditions — Osteoarthritis, Hip; Femoral Neck Fractures; Femur Head Necrosis | interventions — Arthroplasty, Replacement, Hip; Second-Look Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SYMBOL medical devices: Patients undergoing total hip arthroplasty with at least one medical device from the SYMBOL range
  Interventions: Device: Total hip arthroplasty (primary or revision)

INTERVENTIONS:
Device: Total hip arthroplasty (primary or revision) — Total hip arthroplasty with at least one medical device from the SYMBOL range

SUMMARY:
The purpose of this post-market clinical follow up study is to assess the safety and effectiveness of the SYMBOL range of medical devices. The study will evaluate the outcome of Total Hip Arthroplasty using medical devices from SYMBOL range over a period of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years at implantation.
* Patient who will undergo, during the study's period of inclusion, a total hip arthroplasty (primary or revision) with at least one SYMBOL medical device (DEDIENNE Santé).
* Patient informed of his/her participation and willing to participate in the study.
* Patient able to read, write and understand French.

Exclusion Criteria:

* Patient deprived of freedom, under guardianship/curatorship or placed under judicial protection
* Patient unable to follow study procedures.
* Patient who has already been included in the study for a total hip arthroplasty (primary or revision) with at least one SYMBOL medical device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient requiring total hip arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 747 (Estimated)
Dates: Start 2021-09-21 (Actual); Primary Completion 2034-09 (Estimated); Study Completion 2034-09 (Estimated)

PRIMARY OUTCOMES:
Survivorship of 13 individual SYMBOL orthopaedic components | 10 years post-operative
  The survival rate of an orthopaedic implant will be calculated on the basis of the first occurrence of implant revision from any cause.

SECONDARY OUTCOMES:
Survivorship of all individual SYMBOL orthopaedic components | 6 months, 18 months and 5 years post-operative
  The survival rate of an orthopaedic implant will be calculated on the basis of the first occurrence of implant revision from any cause.
Survivorship of the SYMBOL STEM VARA CEM orthopaedic implant. | 10 years post-operative
  The survival rate of an orthopaedic implant will be calculated on the basis of the first occurrence of implant revision from any cause.
Survivorship of the SYMBOL implants by component assembly (acetabular + femoral components) | Through study completion, an average of 10 years
  The survival rate of a combinaison of implant (acetabular + femoral component) will be calculated on the basis of the first occurrence of implant revision from any cause.
Adverse Device Effects. | Through study completion, an average of 10 years
  All adverse device effects occurring from the time of subject enrollment until study termination or study completion including intra-operative adverse events.
  Note: This outcome will also be used for subgroup analyses by component association.
Radiographic assessment - Implant subsidence. | 6 months, 18 months, 5 and 10 years post-operative
  Stem subsidence will be classified based on the following:
  * Stem subsidence < 3mm
  * Stem subsidence between 3 and 5mm
  * Stem subsidence > 5mm
  Note: This outcome will also be used for subgroup analyses by component association.
Radiographic assessment - Osteolysis (granuloma). | 6 months, 18 months, 5 and 10 years post-operative
  Assessment will consider:
  - Presence or absence of osteolysis. If osteolysis is present, impacted areas will be determined according to DeLee and Charnley or Gruen classification.
  Note: This outcome will also be used for subgroup analyses by component association.
Radiographic assessment - Radiolucent lines. | 6 months, 18 months, 5 and 10 years post-operative
  Assessment will consider:
  - Presence or absence of radiolucent lines.
  If radiolucent line is present:
  * Impacted areas will be determined according to DeLee and Charnley or Gruen classification.
  * Type of radiolucent lines will be classified based on the following : < 2mm - regular or > 2mm - irregular.
  Note: This outcome will also be used for subgroup analyses by component association.
Radiographic assessment - Eterotopic ossifications. | 6 months, 18 months, 5 and 10 years post-operative
  Assessment will consider:
  - Presence or absence of eterotopic ossifications. If eterotopic ossification, grade will be specified.
  This outcome will also be measured for subgroup analyses by component association.
Harris Hip Score (or modified Harris Hip Score) at each visit. | Pre-operative, 6 months, 18 months, 5 and 10 years post-operative
  The Harris Hip Score is a joint specific score that consists of 10 items covering domains of pain, function, functional activities, absence of deformity, and hip range of motion.
  Note: This outcome will also be used for subgroup analyses by component association.
Pain intensity (Numeric Rating Scale) | Pre-operative, 6 months, 18 months, 5 and 10 years post-operative
  Numeric Rating scale for pain intensity assessment:
  * Minimum value: 0 (=no pain)
  * Maximum value: 10 (= worst possible pain). (Higher scores mean worst outcome).
  Note: This outcome will also be used for subgroup analyses by component association.
EQ-5D-5L score | Pre-operative, 18 months, 5 and 10 years post-operative
  The EQ-5D-5L score consists of two parts: a descriptive system and a visual analogue scale. The descriptive system is used to describe the subject's health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  The visual analogue scale records the subject's self-rated health on a vertical visual analogue scale.
  Note: This outcome will also be used for subgroup analyses by component association.
Global patient satisfaction | 18 months post-operative
  Ordinal scale for global patient satisfaction assessment:
  - Possible values are: not satisfied/quite satisfied/satisfied/very satisfied ("Very satisfied" is the best possible outcome).
Hip joint patient satisfaction (Numeric Rating Scale) | 5 years and10 years post-operative
  Numeric rating scale : Percentage Scale for Hip Joint Patient Satisfaction Assessment.
  Range of values: from 0 to 100. (100 is the best possible outcome and is equivalent to a normal hip).
  Note: This outcome will also be used for subgroup analyses by component association.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rousseau, Principal Investigator — Clinique Mutualiste Catalane
Locations (9):
- France (9):
  - Hôpital Privé de la Châtaigneraie, Beaumont
  - CH de Marmande - CHIC, Marmande
  - Hôpital Privé du Grand Narbonne, Montredon-des-Corbières
  - Polyclinique Grand Sud, Nîmes
  - Clinique Mutualiste Catalane, Perpignan
  - CH de Péronne, Péronne
  - Clinique Mutualiste, Saint-Etienne
  - Hôpital d'Instruction des Armées Saint-Anne, Toulon
  - Hôpital Robert Schuman - UNEOS, Vantoux